CLINICAL TRIAL: NCT02879708
Title: Effect of Social Accountability on Improving Service Delivery and Outcomes in the Public Sector: a Cluster-Randomized Control Trial in Uttar Pradesh, India
Brief Title: Effect of Social Accountability on Improving Service Delivery and Outcomes in the Public Sector in Uttar Pradesh, India
Acronym: D0168
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: World Bank (Other); University of North Carolina, Chapel Hill (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Manoj Mohanan, Professor, Sanford School of Public Policy, Duke University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-0417; IE-P150365 (Other Grant/Funding Number: World Bank Strategic Impact Evaluation Fund (SIEF))
Record Dates: First submitted 2016-07-25; First posted 2016-08-26 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Health Behavior
Keywords: Social Accountability; Healthcare Quality; Health System Strengthening; Child Health; Childhood pneumonia; Childhood diarrhea
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): 40 (of 120) randomly selected villages receive no intervention
- Information Only (Other): 40 randomly selected villages are assigned to the "information only" arm where households will receive information regarding their rights and entitlements pertaining to healthcare, certain health outcomes specific to their village, as well as health-related activities happening in their village.
  Interventions: Other: Information Only
- Information and Facilitation (Other): The remaining 40 villages will receive similar information as the villages in the Information Only Arm, but will also have facilitators present that ensure the existence of the VHSNC at the village level as well as the occurrence of VHSNC monthly meetings.
  Interventions: Other: Information and Facilitation

INTERVENTIONS:
Other: Information Only — Households will receive information regarding their rights and entitlements pertaining to healthcare, certain health outcomes specific to their village, as well as health-related activities happening in their village (such as the VHSNC meetings and Village Health and Nutrition Days). Information will be disseminated through an initial visit to all households, and from then on either through (1) broadcast messages sent to households via mobile phone, (2) central individuals in the village social network who will be asked to spread that information, or (3) public officials charged with spreading the information throughout the village.
  Arms: Information Only
Other: Information and Facilitation — In addition to the information interventions described above, this intervention will provide trained facilitators to help community members engage in a participatory process with VHSNCs and identify key deficiencies for improvement in health services that most concern community members. The facilitators are trained to help organize meetings and are provided a detailed checklist of activities to be undertaken prior to the the meetings. The three key health workers at the village level (ASHA, ANM, and AWW) report to the local (village level) elected representatives and block level authorities, who receive feedback from the community in the accountability interventions.
  Arms: Information and Facilitation

SUMMARY:
In several low and middle-income countries, Social Accountability (SA) interventions have been introduced as an innovative approach to governance, aiming to improve delivery of public services. These interventions typically include information provision to citizens regarding their rights/entitlements and local provider performance, and additionally, facilitation of community engagement with providers and officials.

The state government of Uttar Pradesh (UP) and the Uttar Pradesh Health Systems Strengthening Project (UPHSSP) have identified 12 districts where the social accountability initiative will be introduced on a priority basis. This study focuses on interventions in 2 of these districts (Sultanpur and Fatehpur), to study mechanisms through which information and collective action lead to improved accountability and outcomes. Within the 2 districts, the study is implemented as a cluster randomized evaluation with 120 villages randomized into 2 treatment arms and one control arm.

This study aims to: (a) measure the causal effect of SA interventions on key outcomes (health status, quality of service); (b) test the effectiveness of social networks based strategies to disseminate information for community engagement; and (c) study individuals' decisions to participate in collective action efforts in the context of social networks and information interventions. In addition to evaluating the impact of the SA interventions, the study aims to generate new knowledge on relative strengths of information seeding strategies, identifying those that maximize the spread of information through the village network, and subsequently estimate peer effects on participation decisions.

DETAILED DESCRIPTION:
The World Bank-supported Uttar Pradesh Health System Strengthening Project (UPHSSP) includes a component that calls for the implementation of social accountability (SA) interventions in UP, which aim to stimulate community action to demand better services, enhance positive health behavior and promote social audits of service delivery and resource allocation. Two key channels through which SA interventions operate are through (a) information provision and (b) fostering community engagement that enables grievance redressal. Prior to the implementation of SA interventions at scale in UP, this study aims to conduct rigorous impact evaluation of key components of SA interventions in order to learn about potential impact in the UP context and to learn about critical implementation issues regarding optimal methods to deliver information in the state with available technology and social networks.

The evaluation's overarching research questions are whether SA interventions in UP improve (1) objective measures of health service quality in practice, (2) village-level satisfaction with health services, and (3) village-level health outcomes. Importantly, the evaluation will seek to identify whether the information provision that is a standard part of social accountability interventions has an independent effect on outcomes that is comparable to the effect of the combined information and community engagement components. The investigators also test the effectiveness of alternative models of delivering information in order to inform implementation of accountability interventions at large scale in public policy settings. Given that the community health workers targeted by the intervention focus on maternal and child health, our measures of health system performance along these three dimensions will also emphasize maternal and child health. Measures of health service quality include availability of services such as immunization and primary care services, distribution of food and nutritional supplementation as recommended in the national nutrition program, and provider absenteeism. Measures of satisfaction with local health services will include process measures including availability of service, waiting time for services and whether or not community members perceive that they are treated by providers with respect as well as general subjective assessments of satisfaction with services. Health outcome measures will include child anthropometrics (weight-for-age and weight-for-height), self-reported morbidity in the preceding two weeks (diarrhea, cough, fever, headache, days of usual activities lost due to illness), and neonatal (0-28 days), infant (under age one), and child (under age five) mortality as well as maternal health indicators such as percentage of facility deliveries among mothers who gave birth in the past year.

Within the 2 study districts (Sultanpur and Fatehpur), in 120 villages that were selected at random, the SA interventions aim to distinguish the effect of provision of information and facilitated engagement of community members, from that of the effect of information alone. The 120 villages are randomized to either a control arm, or one of two treatment arms described below.

TREATMENT ARM 1 - Information & Awareness:

Community members will receive information about their rights, roles and responsibilities of healthcare providers, and also about health-related activities and programs taking place in their village. Importantly, besides assessing the effect of providing information on health service delivery and various health outcomes, our evaluation will also determine how best to provide the information.

Another innovation in this project is to disseminate monthly information about health system related issues using interactive voice response messages (IVRs), phone calls, or home visits to households in the treatment villages. IVRs include a brief message about a health (or health system) indicator, or information regarding upcoming Village Health, Sanitation and Nutrition Committee (VHSNC) meetings or VHNDs, as well as a response option that can be used to collect data on what information households have received and about their participation in VHSNC meetings/VHNDs. These IVRs will be sent out over multiple months to cover approximately 24,000 households in 80 treatment villages each time. During preparatory phase that was conducted in parallel with the baseline survey, detailed data on social networks was collected in each village and identified central individuals in the village.

The investigators will use the data on networks in villages, combined with the information that is disseminated on a monthly basis to econometrically estimate how information dissemination within networks affects awareness and participation in social accountability activities as well as in utilization of health services.

TREATMENT ARM 2 - Information PLUS Community Engagement:

In addition to all the information interventions listed in treatment arm 1, community engagement will be facilitated in Arm 2 villages. The community engagement component aims to enhance the participation of the community in creating social accountability. The intervention will provide trained facilitators to help community members engage in a participatory process with Village Health, Sanitation, and Nutrition Committees (VHSNCs) and identify key deficiencies for improvement in health services that most concern community members. The facilitators are trained to help organize meetings and are provided a detailed checklist of activities that need to be undertaken prior to the day of the meetings such as inviting the block level officers and ensuring that logistics requirements for Village Health and Nutrition Days (VHNDs) are conveyed to VHSNC members in advance of the meetings. The facilitated meetings with healthcare providers and local and block level representatives aim to empower community members to demand better health services and convey these demands more effectively to providers and officials. The three key health workers at the village level (ASHA, ANM, and AWW) report to the local (village level) elected representatives and block level authorities, who receive feedback from the community in the accountability interventions. Moreover, through repeated community meetings village-level health workers are expected to respond to transparency and accountability innovations by improving quality of services delivered to their local constituents resulting in improvements in population health outcomes.

These interventions will focus on services delivered by village-level health workers including those providing primary care and maternal and child health services. The households surveyed in the project will be those with children less than 5 years of age. The interventions will cover and include all population subgroups, castes, and religious minorities in the treatment villages, and also collect data on all of these subgroups.

ELIGIBILITY:
Inclusion Criteria:

* households residing in the villages selected for the evaluation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105000 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Weight-for-height Z scores | 12 months after intervention implementation

SECONDARY OUTCOMES:
Satisfaction with providers - averaged from a rating index and/or constructed by a PCA on the rating index | 12 months after intervention implementation
  Level of satisfaction with local healthcare providers, as estimated by (1) averaging rating scores across a satisfaction index (questions asking the respondent to rate aspects of their last experience with the provider on a scale of 1-5); and/or (2) running a principal components analysis on the same index and taking the first component.
Participation - as measured from self-report | 4 months, measured each month, and at 1 year during endline survey
  household participation in VHSNC meetings and attendance at VHNDs, measured by self-report
U5 mortality rate | 12 months after intervention implementation
  under 5 mortality rates
incidence of diarrhea | 12 months after intervention implementation
duration of diarrhea illness | 12 months after intervention implementation

OTHER OUTCOMES:
Info spread | 4 months, measured each month
  proportion of the village that received/retained information spread through the different info dissemination strategies

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Mohanan, PhD, MSPH, Principal Investigator — Duke University
Locations (1):
- Uttar Pradesh State Institute of Rural Development, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to make the de-identified data set publicly available.

REFERENCES:
- [Background] Ringold, D., Holla, A., Koziol, M., & Srinivasan, S. (2012).